CLINICAL TRIAL: NCT07254507
Title: Evaluation of Lung Ultrasound-Guided Posture Management for Improving Outcomes in Neonatal Ventilator-Associated Pneumonia
Brief Title: Lung Ultrasound-Guided Positioning Strategy for the Prevention of Ventilator-Associated Pneumonia in Neonates
Acronym: LUS-POSforVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huiyi Li (Other)
Responsible Party: Sponsor-Investigator, Huiyi Li, Nurse, Deputy Director of Pediatrics, the Second People's Hospital of Guangdong Province affiliated to Jinan University., Guangdong Second Provincial General Hospital
Organization: Guangdong Second Provincial General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-KY-KZ-266-02; 2024A03J0771 (Other: Guangzhou science and technology plan project)
Record Dates: First submitted 2025-11-15; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia
Keywords: Pulmonary ultrasound; Body position management; Neonatal ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard positioning management (Placebo Comparator): NICU routine nursing
  Interventions: Behavioral: standard positioning management
- LUS-Guided Group (Lung Ultrasound-Guided Positioning) (Experimental): In addition to standard care, LUS assessments were conducted twice daily at fixed time points (08:00 and 18:00) to evaluate regional aeration and guide individualized postural adjustments.
  Interventions: Behavioral: Lung Ultrasound Guided Localization

INTERVENTIONS:
Behavioral: standard positioning management — Infants in the control group had their positions adjusted every two hours, alternating between supine, left lateral, right lateral, and prone positions.The head of the bed should be elevated 15°-30° with the body in a slightly flexed position-hips aligned along the midline, shoulders slightly forward, head centered, and arms free to move. Position adjustments should only be made when vital signs are stable and resuscitation is delayed, or when adjusting the ventilator, administering IV fluids, or managing deep sleep. If heart rate fluctuates more than 20 beats per minute or SpO₂ drops below 90% (excluding airway obstruction), the interval between position adjustments should be extended to 3-4 hours. This group did not undergo ultrasound evaluation.
  Arms: Standard positioning management
Behavioral: Lung Ultrasound Guided Localization — In addition to routine care, two LUS assessments are conducted at fixed times daily (08:00 and 18:00) to guide individualized position adjustments by monitoring regional ventilation.①If unilateral atelectasis or pulmonary edema is detected, the patient should first be maintained in dependent lateral position for approximately 1 hour, then transition to the contralateral or prone position for 3 hours.②For lesions previously managed by the department, the prone position duration is reduced to 1 hour, while supine or lateral positions are extended to 3 hours. ③For posterior lesions, the supine or lateral position should be limited to 1 hour, while the prone position should be extended to 3 hours.④Resume the standard two-hour shift system once the symptoms or edema have subsided.If SpO₂ remains persistently below 90% (excluding operational or feeding disturbances), the respiratory rate increases by more than 20 breaths per minute from baseline, an additional LUS evaluation is required.
  Arms: LUS-Guided Group (Lung Ultrasound-Guided Positioning)

SUMMARY:
This study aims to determine if using lung ultrasound to guide personalized positioning for ventilated newborns is more effective than standard repositioning at preventing ventilator-associated pneumonia.

DETAILED DESCRIPTION:
This research study is testing a new strategy to help prevent Ventilator-Associated Pneumonia(VAP) in newborns who need a breathing machine (mechanical ventilator). VAP is a serious lung infection that can sometimes occur in the hospital.We are using abedside Lung Ultrasound (LUS). This is a safe, painless, and radiation-free imaging tool. It allows doctors to see how well different parts of a baby's lungs are inflated in real-time, much like a "window" into the lungs.Based on the lung ultrasound pictures,our healthcare team will create a personalized positioning plan for the baby (for example, placing them more on their side or on their tummy). The goal is to use gravity to help open up the lungs and drain any fluid, which may lower the risk of infection. We will compare this new method to the standard practice of turning babies every two hours.We believe this personalized,evidence-based care strategy could be more effective in preventing pneumonia. It may potentially help babies get off the breathing machine sooner and reduce their time in the neonatal intensive care unit (NICU).Lung ultrasound is a well-established and safe bedside procedure.This study has been carefully reviewed and approved by the hospital's Ethics Committee. All procedures will be performed by trained doctors and staff, with the baby's safety and comfort as our top priority.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants included term neonates (gestational age 37-42 weeks) who required invasive mechanical ventilation for more than 48 hours.

Exclusion Criteria:

* Exclusion criteria included ①preterm neonates; ② Neonates with early sepsis or previous pneumonia;③ Not suitable for patients with enteral nutrition;④ Newborns requiring mechanical ventilation due to surgery;⑤ There are many infants with congenital abnormalities or suspected chromosomal abnormalities.

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ventilator-associated pneumonia in neonates | From randomization until VAP diagnosis, successful extubation, or death, whichever occurs first, assessed up to 100 days.
  Pneumonia that occurs 48 hours after mechanical ventilation (MV) and 48 hours after extubation is an important type of Hospital-acquired pneumonia (HAP), in which pneumonia that occurs within MV≤4 days is early-onset VAP, and pneumonia that occurs within MV ≥5 days is late-onset VAP.

SECONDARY OUTCOMES:
feeding intolerance in newborns | From the beginning of enteral feeding to the successful establishment of full enteral feeding, discharge or death. The evaluation will last until the end of the study, and the longest evaluation period for each participant is expected to be 100 days.
  Incidence of feeding intolerance at any level (mild+severe)
Pulmonary hemorrhage | From the day of random grouping to the event, discharge or death, whichever comes first. The evaluation lasts for the whole invasive mechanical ventilation period and 24 hours after extubation, and the longest evaluation period is expected to be 100 days
  Incidence of any grade of pulmonary hemorrhage
Pneumothorax | From the day of random grouping to the event, discharge or death, whichever comes first. The evaluation lasts for the whole invasive mechanical ventilation period and 48 hours after extubation, and the longest evaluation period is expected to be 100 days
  Incidence of pneumothorax
new intracranial hemorrhage | From the day of random grouping to the end of discharge or study period, whichever comes first. Routine monitoring will last until the seventh day after birth, and the longest evaluation period is expected to be 120 days.
  The incidence of any new intracranial hemorrhage (including symptomatic and asymptomatic)
Mortality | From the day of random grouping to the end of discharge or study period, whichever comes first. The longest evaluation period is expected to be 120 days.
  Mortality during hospitalization
Duration of invasive mechanical ventilation | Time is counted from invasive ventilation to successful extubation or death. The evaluation will last until the end of the study, and the longest evaluation period for each participant is expected to be 100 days.
  Duration of ventilator use: from start to successful extubation or death.
NICU hospitalization duration | Time is counted from admission to transfer out of NICU or discharge. The evaluation will last until the end of the study, and the longest evaluation period for each participant is expected to be 120 days.
  Time from admission to discharge for hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Guangdong Province affiliated to Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
This study plans to share the collected individual participant data after de-identification.Specifically, it includes: demographic data (gestational age, birth weight, etc.), baseline characteristics, data related to VAP diagnostic criteria, lung ultrasound results, position adjustment records, mechanical ventilation duration, and all primary and secondary endpoint data (feeding intolerance, pulmonary hemorrhage, new intracranial hemorrhage, mortality rate, hospitalization days in NICU, etc.).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be provided within 6 months after the publication of the main results of this study, and the data will be shared for at least 5 years.
Access Criteria: To provide researchers who provide research proposals with rigorous methodology and clear scientific objectives for achieving the research objectives in the approved proposals. It usually includes meta-analysis of individual participant data, verification of results, or exploration of new scientific hypotheses that conform to the original research ethical framework.The proposal should be submitted to: liangzhenyu0823@163.com (please note: please replace this with the official contact email you wish to use).
  To gain access, the applicant needs to sign a data use agreement. The research steering committee of this study will review the scientific value and methodological rigor of the proposal.
URL: https://register.clinicaltrials.gov/prs/beta/studies/S000GENM00000083/protocol/ipdSharing?edit=true

DOCUMENTS (2):
  • Study Protocol (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT07254507/Prot_000.pdf
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT07254507/ICF_001.pdf